CLINICAL TRIAL: NCT06030440
Title: De-Intensification of Postoperative Radiotherapy in Patients with Squamous Cell Carcinoma of the Head and Neck
Acronym: DIREKHT2
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DIREKHT2
Record Dates: First submitted 2023-08-11; First posted 2023-09-11 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-10

CONDITIONS: Squamous Cell Carcinoma of the Oral Cavity; Squamous Cell Carcinoma of the Larynx; Squamous Cell Carcinoma of the Hypopharynx; Squamous Cell Carcinoma of the Oropharynx
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control Arm (Active Comparator): postoperative radiotherapy of the head and neck region according to current standard including elective nodal irradiation
  Interventions: Radiation: RT standard of care
- Investigational Arm (Experimental): postoperative radiotherapy of the head and neck region without elective nodal irradiation
  Interventions: Radiation: Eliminating RT to the elective neck

INTERVENTIONS:
Radiation: Eliminating RT to the elective neck — Reduction of radiation volume by eliminating radiotherapy to the elective neck
  Arms: Investigational Arm
Radiation: RT standard of care — postoperative radiotherapy of the head and neck region according to current standard including elective nodal irradiation
  Arms: Control Arm

SUMMARY:
This randomized, prospective, multicenter phase II/III trial will study the reduction of radiation volume by eliminating radiotherapy (RT) to the elective neck using strictly defined surgical and radio-oncological standards to reduce radiotherapy-related long-term side effects without affecting locoregional control.

DETAILED DESCRIPTION:
This study aims to determine whether it is possible to achieve an individual target volume concept that eliminates elective irradiation of uninvolved lymph drainage areas while maintaining clearly defined surgical standards and using modern imaging and radiation techniques. The aim of this study is to achieve reduced late toxicity without compromising locoregional control.

Patients will be randomized to: either RT to primary tumor region, regions with lymph node metastases and elective nodal irradiation (control arm) or RT to primary tumor region and regions with lymph node metastases without elective nodal irradiation (investigational arm)

A two-stage design was chosen for this purpose.

Phase II:

A randomized phase II study whose primary endpoint is the 1-year percutaneous endoscopic gastrostomy (PEG) tube dependence rate will be performed first.

Phase III:

If the primary endpoint of the phase II study is met and the interim analysis shows no increase in the locoregional recurrence rate in the study/investigational arm, the study will be continued as a phase III study whose primary endpoint is the locoregional control rate.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically proven squamous cell carcinoma of the oral cavity/larynx/oro-or hypopharynx (except glottis cancer (pT1/2pN0))
2. Surgery of primary tumor and neck dissection performed according to predefined surgical standard
3. Indication for postoperative radio(chemo)therapy
4. No lymph node metastases > 6cm
5. Lymph node metastases in not more than 3 lymph node level
6. No distant metastases (cM0)
7. Age ≥ 18 years, no upper age limit
8. Eastern Cooperative Oncology Group (ECOG) ≤ 2
9. Patients who understood protocol contents and are able to behave according to protocol
10. Signed study-specific consent form prior to therapy
11. Start of radiotherapy at least 6 weeks after last tumor-specific surgery (e.g. resection primary tumor, neck dissection, excluded are surgeries according to wound healing complications)

Exclusion Criteria:

1. macroscopic incomplete resection R2
2. Distant metastases (cM1)
3. Radiologically or histologically proven early recurrence after surgery (time frame from surgery to start of radio(chemo)therapy)
4. Lymph node metastases in > 3 lymph node level
5. pregnant or lactating/nursing women
6. fertile patients that are not willing to use highly effective methods of contraception (per institutional standards) during treatment
7. Any condition potentially hampering compliance with the study protocol and follow-up schedule
8. On-treatment participation on other clinical therapeutic trials
9. Prior tumor-specific therapy any other than surgery (like prior radiotherapy in the head and neck region, prior chemo- or immunotherapy (neoadjuvant/induction))
10. Patients who have contraindication for MRI and CT with contrast agent (both)
11. Prior (> 2 months before beginning of radio(chemo)therapy) neck dissection or surgery in the head and neck area affecting lymph drainage
12. History of another primary malignancy except for malignancy treated with curative intent and with no known active disease ≥5 years before diagnosis of head and neck cancer, adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease, adequately treated carcinoma in situ without evidence of disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 508 (Estimated)
Dates: Start 2024-01-26 (Actual); Primary Completion 2031-12 (Estimated); Study Completion 2033-09 (Estimated)

PRIMARY OUTCOMES:
Phase II: 1-year PEG feeding tube dependence rate | PEG-dependent 1 year after radiotherapy
  observe change of PEG-dependence due to different target volumes
Phase III: Time to local relapse | From the date of randomization until the date of observation of local relapse or the date of last observation if no LR occurred, whichever came first (assessed up to 26 months)
  difference between the date of randomization and the date of observation of local relapse (LR), or the date of last observation if no LR occurred (censored observation)

SECONDARY OUTCOMES:
Disease-free survival | up to 26 months
  Disease-free survival
Distant-metastasis-free survival | through study completion, an average of 26 months
  Distant-metastasis-free survival
Overall survival (OS) | up to 26 months
  Overall survival (OS)
Cause of death (tumor-related, not tumor-related) | through study completion, an average of 26 months
  Cause of death (tumor-related, not tumor-related)
Acute toxicity according to Common Terminology Criteria (CTC) version 5.0 | up to 2 months
  Acute toxicity according to CTC version 5.0
Late toxicity according to CTC version 5.0 | up to 24 months
  Late toxicity according to CTC version 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Sarina Müller, PD, Study Director — Universitätsklinikum Erlangen, HNO; Rainer Fietkau, Prof, Principal Investigator — Universitätsklinikum Erlangen, Radiation Oncology
Locations (1):
- Universitätsklinikum Erlangen, Strahlenklinik, Erlangen, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: No